CLINICAL TRIAL: NCT03532659
Title: Impact of Active Video Game Cardiorespiratory, Macro and Microcirculation Function of Adolescents With Overweight: Randomized Intervention Study
Brief Title: Impact of Active Video Game on Cardiorespiratory, Macro and Microcirculation Function of Adolescents With Overweight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Universidade Estadual da Paraíba (Unknown)
Responsible Party: Principal Investigator, Thacira Dantas Almeida Ramos, Doctorate, Professor Fernando Figueira Integral Medicine Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Active video game-1
Record Dates: First submitted 2018-03-15; First posted 2018-05-22 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Overweight and Obesity; Cardiovascular Risk Factor; Physical Activity
Keywords: adolescents; obesity; lung function; microcirculation; intima media thickness
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Intervention Model Description: Intervention with two comparison groups. The control or experimental group will be randomly defined by school
  * "Experimental" group: will perform physical activity through the use of the active videogame associated with a gamification strategy three times a week for 50 minutes for a period of 8 weeks.
  * Control group: there will be no intervention proposal, only used for data comparison.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active video game (Experimental): The adolescents will be submitted to physical activity with active video game for 50 minutes, 3 times a week, for a period of eight weeks. The XBOX360® platform will be used with the Kinect accessory (Microsoft®) and Just Dance will be the selected game. The music used for intervention will be previously selected, including those that can lead to moderate intensity, and assembled in blocks of 10. For each week, a new block and challenges must be elaborated to increase the motivation to carry out the physical activity.
  Interventions: Other: Active video game
- control (No Intervention): A follow-up will be done for eight weeks to compare the variables. The adolescents in this group will be interviewed monthly to detect changes in eating habits and lifestyle.

INTERVENTIONS:
Other: Active video game — Among the 20 municipal schools, two will be selected between those with 298 or more students (corresponding to the third quartile of the number of students per school). Next will be selected the school in which the adolescents will be submitted to intervention, and the students from the other school will be control. The intervention will aim to promote physical exercise through active video game XBOX 360 with Kinect. The game selected will be Just Dance, to allow the participation of up to four students at the same time. In addition, a gamification protocol will be performed to increase the adolescents engagement in the exercise.
  Arms: Active video game

SUMMARY:
This study evaluates the effects of physical exercise through active videogame in the microcirculation, macrocirculation, cardiorespiratory function and physical fitness in overweight adolescents. For that, they will be randomized into two groups, one being a control group and the other intervention group. The randomization will be made by school. The intervention group will perform the physical exercise through the active video game, three times a week, for 50 minutes, during 8 weeks. Reassessments will be performed before and after the intervention to evaluate the outcome variables.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese adolescent
* Students enrolled in public schools

Exclusion Criteria:

* Motor, cognitive or pulmonary limitation
* Genetic syndrome
* Pregnancy
* Use of medication that changes the lipid or glucose profile
* Not being treated for overweight

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Microcirculatory blood flow during rest (RF) | 10 minutes
  Variable measured in perfusion units (PU), obtained during the first five minutes of the microcirculation evaluation protocol by Cutaneous Laser Doppler Flowmetry (LDF).
Maximum blood flow (MF) | 10 minutes
  Peak blood flow during post-occlusive reactive hyperemia (PORH), expressed in perfusion units (PU).
Area of hyperemia | 10 minutes
  Scalar numerical variable corresponding to the geometric area related to the process of reflex hyperemia after the mechanism of arterial occlusion, expressed in perfusion units (PU).
Relationship between peak flow during PORH and resting blood flow. | 10 minutes
  Continuous variable, MF / RF ratio expressed in perfusion units (PU).
PORH index | 10 minutes
  Scalar numerical variable related to reactive hyperemia after the arterial occlusion. mechanism, expressed in perfusion units (PU)
Occlusion area | 10 minutes
  Scalar numerical variable corresponding to the geometric area related to the region without reflex hyperemia after the arterial occlusion mechanism, expressed in perfusion units (PU).
Carotid Intima Media Thickness | 30 minutes
  Variable measured in millimeters, obtained by the maximum value of 3 measurements performed in the right common carotid artery and 3 measurements in the left common carotid artery. Performed with a portable device (General Eletric®, LogicE® model), with a high definition linear transducer.
Femoral Intima Media Thickness | 30 minutes
  Variable measured in millimeters, obtained by the maximum value of 3 measurements made in the right femoral artery and 3 measurements in the left femoral artery. Performed with a portable device (General Eletric®, LogicE® model), with a high definition linear transducer.
Cardiorespiratory Fitness - Maximum oxygen consumption | 10 minutes
  Numerical, continuous, expressed in liters per minute per kilogram (l/mim/kg), obtained indirectly through the 20-meter run test.
Flexibility | 5 minutes
  variable numeric, continuous, expressed in centimeters, obtained through the sit-and-reach test.
Abdominal resistance | 2 minutes
  numerical, continuous variable, expressed in absolute number of abdominal performed in one minute, obtained through the sit-up test.

SECONDARY OUTCOMES:
nutritional status | 10 minutes
  measured weight (kilogram) and height (centimeters) for calculating body mass index, expressed in Kg/m^2.
abdominal adiposity | 5 minutes
  measurement of abdominal circumference with inelastic tape, in centimeters.
Blood Pressure | 15 minutes
  measurement blood pressure (mmHg) through digital tensiometer OMRON.
Lung Function - Forced Expiratory Volume in the first second | 20 minutes
  Evaluated by spirometry, with a computerized ultrasonic portable spirometer, with flow sensor, Easy One® brand, with internal Winspiro Software upgrade version 1.04 for connection to computer. The course will provide the values of Forced Expiratory Volume in the first second expressed in liters (l) and in percentage of the predicted value individually (%pred).
Lung Function - Total Lung Capacity | 20 minutes
  Evaluated by spirometry, with a computerized ultrasonic portable spirometer, with flow sensor, Easy One® brand, with internal Winspiro Software upgrade version 1.04 for connection to computer. The course will provide the values of Total Lung Capacity expressed in liters (l) and in percentage of the predicted value individually (%pred).
Strength of the inspiratory and expiratory muscles | 20 minutes
  Evaluated by digital manovacuometry, through a digital manovacuometer MVD300, will be obtained the measurement of respiratory maximum static pressures, maximum inspiratory pressure regarding inspiratory muscle strength and maximum expiratory pressure regarding the expiratory muscles. Both will be expressed in cmH2O.
Fasting blood glucose | 5 minutes
  Continuous numeric variable expressed in mg/dL.
C-reactive protein | 5 minutes
  Continuous numeric variable expressed in mg/dL.
Total cholesterol | 5 minutes
  Continuous numeric variable expressed in mg/dL.
High density lipoprotein (HDL) cholesterol High density lipoprotein (HDL) cholesterol | 5 minutes
  Continuous numeric variable expressed in mg/dL.
Triglycerides | 5 minutes
  Continuous numeric variable expressed in mg/dL.
Glycated hemoglobin A1c | 5 minutes
  Continuous numeric variable expressed in percentage (%).
Low density lipoprotein (LDL) cholesterol | 5 minutes
  Continuous numeric variable obtained by the Friedewald formula= Cholesterol Total - (High Density Lipoprotein + Triglyderides/5), expressed in mg/dL.
Quality of life assessment | 20 minutes
  application of validated questionnaire
Food consumption | 20 minutes
  application of validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Carla CM Medeiros, PhD, Principal Investigator — Universidade Estadual da Paraíba; João Guilherme B Alves, PhD, Study Director — Professor Fernando Figueira Integral Medicine Institute
Locations (2):
- Brazil (2):
  - Escola Municipal de Ensino Fundamental Governador Antônio Mariz, Campina Grande, Paraíba
  - Escola Municipal de Ensino Fundamental Tiradentes, Campina Grande, Paraíba